CLINICAL TRIAL: NCT03582488
Title: Longitudinal Imaging Biomarkers of Disease Progression in DLB
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Kejal Kantarci (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Kejal Kantarci, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-011339; U01NS100620 (NIH)
Record Dates: First submitted 2018-06-21; First posted 2018-07-11 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Lewy Body Disease
MeSH Terms: conditions — Lewy Body Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dementia with Lewy Bodies (Experimental): 18F-Flortaucipir and 11C-Pittsburgh compound-B radioligands will be used for experimental PET imaging of beta-amyloid and neurofibrillary tau pathology
  Interventions: Drug: 18F-Flortaucipir

INTERVENTIONS:
Drug: 18F-Flortaucipir — Radioligands for PET imaging of beta-amyloid and neurofibrillary tangle tau pathology
  Other Names: 11C- Pittsburgh Compound-B

SUMMARY:
The Researchers are trying to determine the paths of change in imaging biomarkers of Dementia with Lewy bodies (DLB) and their associations with rate of cognitive and functional decline.

DETAILED DESCRIPTION:
The proposed project will enroll 90 subjects with probable DLB, 60 from Mayo Clinic Rochester (MCR) and 30 from Mayo Clinic Jacksonville (MCJ). Additionally, 45 controls will be enrolled, 30 from MCR and 15 from MCJ. We will obtain up to six assessments in each subject over the 5 years of the study, baseline, six month and annually thereafter. We will follow these cohorts with clinical and biospecimen data collection annually and once at six months, and CSF collection annually within the guidelines of the Parkinson's Disease Biomarker's Program (PDBP). Clinical neuroimaging will be performed annually and include: a) dopamine transporter imaging with Ioflupane (123I) SPECT (DaTscan) as the biomarker of LBD-related loss of dopaminergic activity, b) structural MRI AD- signature atrophy as the biomarker of AD-related neurodegeneration, c) β-amyloid (Aβ) deposition on PET as the biomarker of Aβ pathology. In patients from the MCR site, we will investigate AV-1451 PET. Since the specificity of AV-1451 PET is not established for tau deposition in DLB, we will investigate this biomarker in a subset of DLB patients to determine the pattern of AV-1451 uptake compared to clinically normal controls, and its association with atrophy, Aβ load and clinical disease progression in DLB.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable DLB, at least 18 years of age, reliable informant who personally speaks with or sees the participant at least weekly, sufficiently fluent in English, must be willing and able to consent to the protocol and undergo up to 6 visits over 5 years, willing and able to undergo neuropsychological testing and no contraindication to MRI imaging.

Exclusion Criteria:

* Presence of another neurologic disorder which could impact findings, such as multiple sclerosis, brain tumors, etc., unwilling to return for follow-up yearly and undergo neuropsychological testing and MR imaging, if undergoing Tau imaging cannot have QT Prolongation, do not have a reliable informant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rate of change in 18F-Flortaucipir PET imaging and Pittsburgh compound-B PET imaging | Will be assessed 3 times annually over at least three years
  Cortical 18F-Flortaucipir and Global cortical Pittsburgh compound-B uptake will be measured in each participant over three years

CONTACTS AND LOCATIONS:
Overall Officials: Kejal Kantarci, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials